CLINICAL TRIAL: NCT00003439
Title: A Phase I Dose-Escalating Study of Recombinant Human Interleukin-12 (NSC # 672423) Administered by Intraperitoneal Infusion in Refractory Advanced Stage Ovarian Cancer and Other Abdominal Carcinomatosis
Brief Title: Interleukin-12 in Treating Patients With Refractory Advanced-Stage Ovarian Cancer or Abdominal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02272; PCI-98-031; PCI-MWH-97-039; NCI-T97-0031; CDR0000066467 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2007-04

CONDITIONS: Cancer
Keywords: stage IV colon cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent pancreatic cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage IV anal cancer; recurrent anal cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; advanced adult primary liver cancer; recurrent adult primary liver cancer; stage IV endometrial carcinoma; recurrent endometrial carcinoma; small intestine adenocarcinoma; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; stage IV prostate cancer; recurrent prostate cancer; fallopian tube cancer; primary peritoneal cavity cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Anus Neoplasms; Carcinoma, Ovarian Epithelial; Carcinoma, Hepatocellular; Endometrial Neoplasms; Gallbladder Neoplasms; Bile Duct Neoplasms; Prostatic Neoplasms; Fallopian Tube Neoplasms | interventions — Interleukin-12 Subunit p35

ARMS (1):
- Arm I (Experimental): Cohorts of 3-6 patients each receive escalating doses of intraperitoneal recombinant human interleukin-12 (rhIL-12) administered weekly for 9 weeks. If a patient tolerates rhIL-12 and shows evidence of objective response or stable disease, patient may receive up to 9 additional weeks of treatment. Treatment continues in the absence of unacceptable toxicity or disease progression. Dose escalation continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which no more than 1 of 6 patients experiences dose limiting toxicity.
  Interventions: Biological: recombinant interleukin-12

INTERVENTIONS:
Biological: recombinant interleukin-12

SUMMARY:
Phase I trial to study the effectiveness of interleukin-12 in treating patients with refractory ovarian or abdominal cancers. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a persons's white blood cells to kill cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Assess the safety and maximum tolerated dose of recombinant human interleukin-12 (rhIL-12) administered by intraperitoneal infusion in patients with chemotherapy refractory advanced ovarian cancer and other diffuse abdominal carcinomatosis.

II. Determine the immunopharmacologic profile of rhIL-12 in this patient population.

III. Evaluate the biologic response in selected patients to rhIL-12 administered through intraperitoneal infusions.

OUTLINE: This is a dose escalation, multicenter study.

Cohorts of 3-6 patients each receive escalating doses of intraperitoneal recombinant human interleukin-12 (rhIL-12) administered weekly for 9 weeks. If a patient tolerates rhIL-12 and shows evidence of objective response or stable disease, patient may receive up to 9 additional weeks of treatment. Treatment continues in the absence of unacceptable toxicity or disease progression. Dose escalation continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which no more than 1 of 6 patients experiences dose limiting toxicity.

All patients are followed for survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed intraabdominal cancer
* Diffuse abdominal carcinomatosis Chemotherapy refractory advanced stage ovarian cancer
* Measurable disease
* Residual, recurrent, or metastatic disease beyond the scope of standard curative therapy
* Extension of disease to sites distant to the peritoneal cavity allowed Retroperitoneal lymphadenopathy allowed as long as there is evaluable intraabdominal disease
* No history of progressive brain metastases

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: Karnofsky 70-100%
* Hemoglobin greater than 9 g/dL
* WBC greater than 3,000/mm3
* Platelet count greater than 100,000/mm3
* Bilirubin less than 2.0 mg/dL
* ALT less than 100 U/L
* Creatinine clearance greater than 60 mL/min
* Normal electrocardiogram
* No recent history of cardiac ischemia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Hepatitis B negative
* No evidence of clinical immunodeficiency syndromes or immunodeficiency associated diseases
* No history of autoimmune disease
* No concurrent major illness
* No serious infection requiring intravenous antibiotics
* No active peptic ulcer disease
* Must have free flow of fluid into the peritoneal space
* No leakage from the catheter exit site

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior biologic therapy (6 weeks for interleukin-2)
* No prior recombinant human interleukin-12
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No concurrent systemic chemotherapy
* No concurrent systemic corticosteroids
* No prior radiation therapy to the whole abdomen
* No concurrent radiotherapy
* At least 3 weeks since prior exposure to any investigational drug
* No concurrent investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1998-08; Primary Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Edwards, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States